CLINICAL TRIAL: NCT06835231
Title: Broncho-vascular 'Lung Sparing' Reconstructions and Pneumonectomies in Patients With Non-small Cell Lung Cancer (Nsclc): Short-/Medium-term Results and Quality of Life
Brief Title: Broncho-Vascular Lung Sparing Reconstructions and Pneumonectomies in Patients With Non Small Cell Lung Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: SP2021
Record Dates: First submitted 2024-11-28; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-10

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to evaluate the medium- to long-term results of patients operated with bronchial and/or vascular sleeves. We will also evaluate the differences in terms of complications and medium-term results with patients undergoing pneumonectomy.

DETAILED DESCRIPTION:
Many studies have confirmed the validity in functional and prognostic terms of resections lung 'lung-sparing' or 'broncho-vascular sleeve' resections), i.e. with sparing of lung parenchyma.

This concept is applicable to small peripheral neoplasms for which there is increasing use of segmental resections instead of lobar resections, but above all - and this is the subject of the present study - for larger neoplasms and/or neoplasms that develop in the proximity of hilar structures with involvement of vascular-bronchial afferents. They are widely described in the literature as bronchial and vascular reconstruction techniques that allow both the preservation of a significant portion of lung parenchyma and consensually guarantee the surgical procedure's oncological radicality.

In addition to the preservation of a functionally valid and effective portion of the lung, with the unquestionable benefits in terms of quality of life for the patient, this type of technique surgical technique with reconstruction offers an additional advantage, making it possible to avoid sacrificing sacrifice of the entire lung (pneumonectomy procedure), an operation that has a considerably higher morbidity and mortality rate.

However, these techniques can also be associated with complications, some of them specific and inherent to (a) the bronchial anastomosis (which may go into dehiscence or stenosis) or b) arterial plastics (in its different forms and with different types of complications); finally, they are procedures that may entail technical surgical difficulties not negligible and are for this reason usually the prerogative of high-volume thoracic surgery centres.

high-volume thoracic surgery centres.

The scientific literature has often focused on long-term oncological outcomes, many studies are available in this regard. In contrast, fewer studies have focused on the short-to-medium-term results (peri-operative period and period within <5aa) and the quality of life of life experienced by the patient after surgery. For example, the development of stenosis cicatricial stenosis of the bronchial anastomosis as well as other technique-specific issues (effectiveness of pulmonary vascular axis reconstruction) has only rarely been explored in detail.

The aim of this study is to examine the characteristics and risk factors of patients undergoing sleeve surgery who subsequently developed anastomosis stenosis or technical complications in a broader sense and the results in terms of prognosis from an oncological point of view.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 years or older (>18 years) who underwent sleeve lung resection in the period between 01.01.2010 to 31.12.2020 for NSCLC.
* For the group undergoing pneumonectomy patients aged 18 years or older (>18 years) undergoing pneumonectomy for NSCLC will be included in the same period (01.01.2010 and 31.12.2020).
* Informed consent for participation in the study.

Exclusion Criteria:

* Other neoplasm treated with chemotherapy in the 3 years prior to lung resection surgery.
* Pathologic involvement N3 or stage IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing sleeve lobectomy or pneumonectomy at the O.U. of Thoracic Surgery of the IRCCS Azienda Ospedaliero Universitaria di Bologna from 01.01.2010 to 31.12.2020.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-09-11 (Estimated); Study Completion 2025-11-11 (Estimated)

PRIMARY OUTCOMES:
Complication rate | through study completion, an average of 18 months
  Rate of postoperative complication
Overall Survival | through study completion, an average of 18 months
  Overall Survival, from the date of surgery to the latest follow up or death
Disease-Free Survival | through study completion, an average of 18 months
  Disease Free Survival, from the date of surgery to the first appearance of local, regional and/or distant recurrence

SECONDARY OUTCOMES:
Early postoperative mortality | 30 and 90 days from the day of surgery
  Mortality rate at 30 and 90 days from the day of surgery
Re-hospitalization | 30 days from the date of discharge
  Rate of rehospitalization in the first 30 days after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Bertoglio, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero Universitaria di Bologna, Bologna, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: Undecided